CLINICAL TRIAL: NCT01866072
Title: A Prospective Evaluation of the Role of Transient Elastography (Fibroscan) in Differentiating Patients of Acute Severe Viral Hepatitis and Acute on Chronic Liver Failure
Brief Title: Evaluation of Role of Transient Elastography (Fibroscan) in Differentiating Patients of Acute Severe Viral Hepatitis and Acute on Chronic Liver Failure
Acronym: ACLF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Dr. Praveen Shrama, Associate professor & Consultant, Sir Ganga Ram Hospital
Other Study IDs: EC/01/13/455
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Acute Severe Viral Hepatitis; Acute on Chronic Liver Failure
Keywords: ACLF; AVH; Fibroscan; Transient elastography
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AVH: AVH: Patients with Acute Viral Hepatitis
- ACLF: ACLF: Patients with Acute on Chronic Liver Failure

SUMMARY:
Transient elastography is novel non-invasive method for assessment of hepatic fibrosis in patients with chronic liver disease, by measuring liver stiffness. Transient elastography is a user friendly technique that can be easily performed at bedside or in outpatient clinic with immediate results and good reproducibility.

Liver stiffness values ranges from 2.5 to 75 kPa with lower values <6kPa suggest no fibrosis where as higher values above 14kPa suggests cirrhosis. In the present study the investigators hypothesis that the investigators can differentiate ACLF and acute severe viral hepatitis based on fibroscan as patients with underlying fibrosis with superadded inflammation would have higher fibroscan value than when patient have only inflammation with no underlying fibrosis and hence the investigators can avoid unnecessary test in such subgroup.

DETAILED DESCRIPTION:
Transient elastography is a novel non-invasive method that for the assessment of hepatic fibrosis in patients with chronic liver diseases, by measuring liver stiffness.

Acute on chronic liver failure: acute hepatic insult manifesting as jaundice and coagulopathy, complicated within 4 weeks by ascites and/or encephalopathy in patients with previously diagnosed or undiagnosed chronic liver disease.

Acute severe hepatitis: Acute severe hepatitis which is characterized by serum bilirubin > or = 10.0 mg/dL and international normalized ratio (INR) > or = 1.5.

Patients with acute severe viral hepatitis or acute on chronic liver failure will be enrolled in this prospective study after taking informed written consent. All patients will be evaluated at baseline as per standard protocol which include evaluation of etiology of disease and tests to exclude underlying liver disease which includes ultrasound/computed tomography and if necessary upper gastrointestinal endoscopy and liver biopsy if imaging shows any signs of underlying liver disease. the patients will be followed up for 1 month, all patients will undergo Fibroscan at the time of admission and thereafter at 1week and 4th week .

ELIGIBILITY:
Inclusion Criteria:

* Patient's age 18-70years.
* Patients with a diagnosis of acute severe viral hepatitis or acute on chronic liver failure.
* Patients willing for informed consent and follow up for 1 month.

Exclusion Criteria:

* Patients with gross ascites, hepatic encephalopathy.
* Patient fail to give written consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute severe viral hepatitis or acute on chronic liver failure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-11 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Fibroscan value at admission | 1st Day
  The patient enrolled will undergo fibroscan procedure and baseline fibroscan values will be measured at the time of admission.

SECONDARY OUTCOMES:
Fibroscan value at week 1 | 1st week
  2nd fibroscan will be done at week 1 from date of admission.
Fibroscan value at week 4 | 4th week
  3rd Fibroscan will be done at 4th week from date of admission.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Arora, M.D, Principal Investigator — Deptartment of gastroenterology & hepatology, Sir Ganga Ram Hospital; Praveen Sharma, M.D, Principal Investigator — Department of Gatroenterology & Hepatology, Sir Gnaga Ram Hospital
Locations (1):
- Department of Gastroenterology & Hepatology, Sir Ganga Ram Hospital, New Delhi, New Delhi, India

REFERENCES:
- [Background] Roulot D, Czernichow S, Le Clesiau H, Costes JL, Vergnaud AC, Beaugrand M. Liver stiffness values in apparently healthy subjects: influence of gender and metabolic syndrome. J Hepatol. 2008 Apr;48(4):606-13. doi: 10.1016/j.jhep.2007.11.020. Epub 2008 Jan 3. PMID 18222014
- [Background] Kumar M, Sharma P, Garg H, Kumar R, Bhatia V, Sarin SK. Transient elastographic evaluation in adult subjects without overt liver disease: influence of alanine aminotransferase levels. J Gastroenterol Hepatol. 2011 Aug;26(8):1318-25. doi: 10.1111/j.1440-1746.2011.06736.x. PMID 21443658
- [Background] de Ledinghen V, Vergniol J. Transient elastography for the diagnosis of liver fibrosis. Expert Rev Med Devices. 2010 Nov;7(6):811-23. doi: 10.1586/erd.10.46. PMID 21050091
- [Background] Castera L, Forns X, Alberti A. Non-invasive evaluation of liver fibrosis using transient elastography. J Hepatol. 2008 May;48(5):835-47. doi: 10.1016/j.jhep.2008.02.008. Epub 2008 Feb 26. PMID 18334275
- [Background] Garg H, Kumar A, Garg V, Sharma P, Sharma BC, Sarin SK. Clinical profile and predictors of mortality in patients of acute-on-chronic liver failure. Dig Liver Dis. 2012 Feb;44(2):166-71. doi: 10.1016/j.dld.2011.08.029. Epub 2011 Oct 5. PMID 21978580
- [Background] McDONOUGH PG, Tho PT, Byrd JR. Twins discordant for 46,XX gonadal dysgenesis. Fertil Steril. 1977 Mar;28(3):251-2. doi: 10.1016/s0015-0282(16)42434-9. PMID 557003
- [Background] Arena U, Vizzutti F, Corti G, Ambu S, Stasi C, Bresci S, Moscarella S, Boddi V, Petrarca A, Laffi G, Marra F, Pinzani M. Acute viral hepatitis increases liver stiffness values measured by transient elastography. Hepatology. 2008 Feb;47(2):380-4. doi: 10.1002/hep.22007. PMID 18095306
- [Background] Kumar M, Satapathy S, Monga R, Das K, Hissar S, Pande C, Sharma BC, Sarin SK. A randomized controlled trial of lamivudine to treat acute hepatitis B. Hepatology. 2007 Jan;45(1):97-101. doi: 10.1002/hep.21486. PMID 17187417